CLINICAL TRIAL: NCT01039753
Title: Analysis of Clinical Outcomes in Patients Undergoing Acute Dialysis Therapy at Intensive Care Units
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yung-Ming Chen, National Taiwan University Hospital
Other Study IDs: 200912015R
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; renal replacement therapy; biomarkers
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collect serum and urine sample for biomarkers at the following timing: start date of renal replacement therapy, discontinuation date of renal replacement therapy, 7 days after discontinuation date of renal replacement therapy. 10ml blood and 10ml urine will be collected at each sampling
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute kidney injury is more frequent and the mortality rate would be as high as 50-60% when the renal replacement therapy was needed. Many studies about the timing of start and discontinuation of dialysis, dialysis dose, dialyzer, anticoagulation and dialysates were initiated but the results were still controversial. In addition, more new biomarkers were found to predict the outcome of acute kidney injury and these biomarkers may play an important role for the dilemma of aforementioned studies.

This observational prospective study has two objectives:

1. To find the predictors of outcome for the acute kidney injury with renal replacement therapy and determine the appropriate method.
2. To find the relationship between new biomarkers and acute kidney injury and determine whether it can be a factor for the monitor of the response of the renal replacement therapy.

DETAILED DESCRIPTION:
Background:

Acute kidney injury is more frequent than before and the incidence rate was about 35-50% in hospital. The mortality rate would be as high as 50-60% when the renal replacement therapy was needed. Many studies about the timing of start and discontinuation of dialysis, dialysis dose, dialyzer, anticoagulation and dialysates were initiated but the results were still controversial. In addition, more new biomarkers were found to predict the outcome of acute kidney injury and these biomarkers may play an important role for the dilemma of aforementioned studies

Objectives:

1. To find the predictors of outcome for the acute kidney injury with renal replacement therapy and determine the appropriate method of renal replacement therapy for acute kidney injury
2. To find the relationship between new biomarkers and acute kidney injury and determine whether it can be a factor for the monitor of the response of the renal replacement therapy.

Methods:

1. Study duration: 2010/01/01 to 2011/6/30
2. Patient eligibility : over 18 years-old and admitted to medical intensive care units of National Taiwan University Hospital
3. A prospective study to collect the parameters including underlying diseases, vital signs, biochemistry data, urine output, disease severity scores, dialysis timing, dialysis dose, dialyzer, anticoagulation agents
4. Collect serum and urine sample for biomarkers if patient agree

Statistics:

Normally distributed variables are expressed as means ± SDs. Statistical significance is set at P<0.05. All statistical analyses are performed with SAS statistical software. Comparisons between two groups are assessed with the student's unpaired t test and Mann-Whitney test. Differences between more than two groups are analyzed by ANOVA (ANOVA) using one-way ANOVA. Survival analyses are made with the Kaplan-Meier survival curve and the Cox proportional hazard model.

Keywords : acute kidney injury, renal replacement therapy, biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years-old and admitted to intensive care units of National Taiwan University Hospital

Exclusion Criteria:

* End stage renal disease
* Terminal disease with estimated life span shorter than 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years-old and admitted to intensive care units of National Taiwan University Hospital
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan